CLINICAL TRIAL: NCT04823377
Title: Impact of a Process Optimizing the Decision to Continue or Stop Cancer Treatments in Patients With Advanced Non-small Cell Lung Cancer.
Acronym: PACT-01
Status: Active, not recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Institut Curie (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Supportive Care
Other Study IDs: IC 2020-05
Record Dates: First submitted 2021-03-29; First posted 2021-03-30 (Actual); Last update posted 2025-11-28 (Actual); Status verified 2025-11

CONDITIONS: Carcinoma, Non-Small-Cell Lung; Advanced Cancer
Keywords: cancer therapy; last days of life; optimization device
MeSH Terms: conditions — Carcinoma, Non-Small-Cell Lung

STUDY DESIGN:
Intervention Model Description: In this prospective comparative study, the rate of systemic oncological treatment during the last month of life will be measured consecutively, over a period of usual management, followed by a period of systematic application of a process of optimization of the medical decision.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Period A: Usual management (Other): Period of end-of-life care as usual
  Interventions: Other: Usual care
- Period B: Process of optimization of the medical decision (Other): Period of systematic and iterative use of a device for optimizing the decision to continue an anti-cancer treatment.
  Interventions: Other: Optimization of the medical decision

INTERVENTIONS:
Other: Usual care — Patients receiving systemic anticancer treatment in their last days of life
  Arms: Period A: Usual management
Other: Optimization of the medical decision — Impact of the use of an optimization device of the decision of cancer treatment on aggressiveness of end of life care
  Arms: Period B: Process of optimization of the medical decision

SUMMARY:
Sequential comparative prospective interventional study evaluating the impact of the use of an optimization device of the decision of cancer treatment on aggressiveness of end of life care. Comparison between a first period, period (A), of care as usual and a second period, period (B), of systematic and iterative use of a device for optimizing the decision to continue an anti-cancer treatment.

DETAILED DESCRIPTION:
We propose to study the optimization of this decision process in an advanced Non-Small-Cell Lung Carcinoma (NSCLC) population, with a Performance Status (PS) ≥ 2 (median survival of approximately 3 months) piloting iteratively (before each decision to continue treatment) a process consisting of an evaluation framework (30 items to be answered by the oncologist with the patient), consolidating:

1. clinical parameters;
2. doctors' expectations regarding the continuation of anticancer treatment;
3. patient expectations and preferences;
4. the possibility of referring the patient to a supportive care specialist and strengthening home care.

The process triggers a dialogue between the patient and the oncologist, based on facts and seeks objectivity, ultimately allowing a shared decision.

In this prospective comparative study, the rate of systemic oncological treatment during the last month of life will be measured consecutively, over a period of usual management, followed by a period of systematic application of a process of optimization of the medical decision.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically or cytologically proven non-small-cell lung carcinoma (NSCLC) including NSCLC with oncogene addiction.
2. Stage IV or IIB/IIIC non irradiable (8th classification TNM, UICC 2015)
3. Patient having completed at least one line of chemotherapy in the context of metastatic disease (or in the context of locoregional disease if the last chemotherapy was less than 6 months ago).
4. ECOG Performance Status ≥ 2.
5. Age ≥ 18.
6. Written informed consent.
7. Patient capable, according to the investigator, to comply with the requirements of the study.

Exclusion Criteria:

1. Small Cell Lung Cancer (including mixed forms).
2. Patient with NSCLC for whom a decision has already been made to permanently discontinue all systemic cancer treatment.
3. Impossible follow up for geographical, social or psychological reason.
4. Inability to answer a questionnaire (language or neurological barrier).
5. Patient under guardianship.
6. Patient being treated in a therapeutic trial.
7. Patient not covered by social security. -

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 364 (Estimated)
Dates: Start 2021-09-24 (Actual); Primary Completion 2026-09-23 (Estimated); Study Completion 2027-09-23 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients receiving systemic anticancer treatment in their last days of life | 24 months
  Comparison of the percentage of patients receiving systemic anticancer treatment in their last 30 days of life during each period

SECONDARY OUTCOMES:
Percentage of chemotherapy | 24 months
  Percentage of chemotherapy (IV, oral) administered in the last 60, 30 and 14 days of life,
Number of emergency room visits | 24 months
  Percentage of patients visiting emergency room visits more than once and of unplanned hospitalizations and intensive care admission in the last month of life.
Percentage of initiation of a new line of chemotherapy | 24 months
  Percentage of initiation of a new line of chemotherapy (IV, oral) in the last month of life
Percentage of immunotherapy and of Tyrosine kinase inhibitor | 24 months
  Percentage of immunotherapy and of Tyrosine kinase inhibitor in the last 60, 30 and 14 days of life.
Percentage of initiation of Tyrosine kinase inhibitor or immunotherapy | 24 months
  Percentage of initiation of Tyrosine kinase inhibitor or immunotherapy in the last month of life.
Use of supportive care | 24 months
  Frequency and precocity of use of supportive care.
Overall survival (OS) | 24 months
  Overall survival (OS) defined as the time from the date of consent to the date of death due to any cause.
Quality of life using QLQ-C15-PAL EORTC (European Organization for Research and Treatment of Cancer) and anxiety with HAD (Hospital Anxiety and Depression) questionnaire | 24 months
  The quality of Life in palliative cancer care patients will be collected with QLQ-C15-PAL EORTC scale and anxiety will be mesured with HAD scale.

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Ange MASSIANI, MD, Principal Investigator — Institut Curie
Locations (25):
- France (25):
  - CH Abbeville, Abbeville
  - CH du Pays d'Aix, Aix-en-Provence
  - CHU Amiens - Hôpital Sud, Amiens
  - CHU Angers, Angers
  - CHR Metz-Thionville - Hôpital de Mercy, Ars-Laquenexy
  - CH Henri Duffaut Avignon, Avignon
  - Institut Sainte-Catherine, Avignon
  - AP-HP Ambroise Paré, Boulogne-Billancourt
  - CHI de Compiègne-Noyon, Compiègne
  - CHU Sud Francilien, Corbeil-Essonnes
  - Clinique des Cèdres, Cornebarrieu
  - CH Intercommunal de Créteil, Créteil
  - CGFL, Dijon
  - CHU Grenoble Alpes, Grenoble
  - CHD Vendée, La Roche-sur-Yon
  - CHRU Lille, Lille
  - Centre Léon Bérard, Lyon
  - Institut Curie, Paris
  - AP-HP Cochin, Paris
  - AP-HP Bichat, Paris
  - AP-HP Tenon, Paris
  - Institut Curie, Saint-Cloud
  - CH Saint-Malo, St-Malo
  - Hôpital Foch, Suresnes
  - Clinique Tessier, Valenciennes

IPD SHARING:
Plan to Share IPD: Yes
Sponsor will share de-identified data sets Documents generated under the project will be disseminated in accordance with Institut Curie policies.
Supporting Information: Study Protocol, SAP
Time Frame: Data requests can be submitted starting 9 months after last article publication and will be made accessible for up to 12 months.
Access Criteria: Access to trial individual participant data can be requested by qualified researchers engaging in independent scientific research, and will be provided following review and approval of a research proposal and Statistical Analysis Plan (SAP) and execution of a data sharing agreement (DSA).